CLINICAL TRIAL: NCT00346359
Title: Conditioning For Hematopoietic Cell Transplantation With Fludarabine Plus Targeted IV Busulfan and GVHD Prophylaxis With Thymoglobulin, Tacrolimus and Methotrexate in Patients With Myeloid Malignancies
Brief Title: Fludarabine and Busulfan Followed by Donor Peripheral Stem Cell Transplant and Antithymocyte Globulin, Tacrolimus, and Methotrexate in Treating Patients With Myeloid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 2041.00; FHCRC-2041.00; GEMZYME-FHCRC-2041.00; CDR0000488969 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: graft versus host disease; chronic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia; chronic myelomonocytic leukemia; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; secondary acute myeloid leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic neutrophilic leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Chronic-Phase; Blast Crisis; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Leukemia, Myelomonocytic, Juvenile; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Congenital Abnormalities | interventions — Antilymphocyte Serum; Busulfan; fludarabine phosphate; Methotrexate; Tacrolimus; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: fludarabine phosphate
Drug: methotrexate
Drug: tacrolimus
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine and busulfan, before a donor peripheral stem cell transplant helps stop the growth of abnormal and cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining abnormal or cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving antithymocyte globulin, tacrolimus, and methotrexate before or after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving fludarabine together with busulfan followed by donor peripheral stem cell transplant and antithymocyte globulin, tacrolimus, and methotrexate works in treating patients with myeloid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the incidence and severity of acute graft-versus-host disease (GVHD) in patients with myeloid malignancies treated with conditioning regimen comprising fludarabine phosphate and busulfan followed by allogeneic peripheral blood stem cell transplantation and GVHD prophylaxis comprising antithymocyte globulin, tacrolimus, and methotrexate.
* Determine the incidence of donor engraftment in patients treated with this regimen.

Secondary

* Determine the pharmacokinetics of IV busulfan, including interdose variability and evaluation of a limited sampling strategy, in these patients.
* Determine the pharmacokinetics of antithymocyte globulin in these patients.
* Determine the pharmacokinetics of fludarabine phosphate and its effect on lymphocytes in these patients.
* Determine the incidence of specific toxic effects ≥ grade 3 in patients treated with this regimen.
* Determine the incidence and severity of chronic GVHD in these patients.
* Determine the incidence of nonrelapsing mortality at 100 days and at 1 year after transplantation in these patients.
* Determine the incidence of relapse in these patients.
* Determine relapse-free survival of these patients.
* Determine the incidence of Epstein-Barr virus activation in these patients.

OUTLINE:

* Conditioning regimen: Patients receive fludarabine phosphate IV over 30 minutes on days -6 to -2 and busulfan IV over 3 hours on days -5 to -2. Prior to the conditioning regimen, patients whose cerebrospinal fluid is positive for malignant cells receive intrathecal methotrexate or cranial irradiation for CNS prophylaxis.
* Allogeneic peripheral blood stem cell (PBSC) transplantation: Patients receive filgrastim (G-CSF)-mobilized allogeneic PBSCs IV on day 0.
* Graft-versus-host disease prophylaxis: Patients receive antithymocyte globulin IV over at least 10 hours on days -3 to -1. They also receive tacrolimus orally twice daily or IV continuously beginning on day -1 and continuing until up to day 55, followed by a taper until day 180 in the absence of graft-versus-host disease. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

After completion of study treatment, patients are followed annually.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following myeloid malignancies:

  * Chronic myelogenous leukemia meeting 1 of the following criteria:

    * Chronic phase
    * Accelerated phase
    * Treated blast phase
  * Acute myeloid leukemia meeting 1 of the following criteria:

    * In remission
    * In early relapse, defined as < 10% marrow blasts
  * Myelodysplastic syndromes, including all risk groups
  * Other myeloproliferative disorders
* HLA-A, -B, -C, -DRB1, and -DQB1 matched related or unrelated donor available

PATIENT CHARACTERISTICS:

* No other disease that would severely limit life expectancy
* AST ≤ 2 times normal
* Creatinine ≤ 2 times normal OR creatinine clearance ≥ 60 mL/min
* No cardiac insufficiency requiring treatment
* No symptomatic coronary artery disease
* PO_2 ≥ 70 mm Hg AND DLCO ≥ 70% of predicted OR PO _2 ≥ 80 mm Hg AND DLCO ≥ 60% of predicted
* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No post-transplantation growth factor during methotrexate administration

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-03; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of acute graft-versus-host disease (GVHD)
Incidence of donor engraftment

SECONDARY OUTCOMES:
Pharmacokinetics of IV busulfan including interdose variability and evaluation of a limited sampling strategy
Pharmacokinetics of antithymocyte globulin
Pharmacokinetics of fludarabine phosphate and its effect on lymphocytes
Incidence of specific toxic effects ≥ grade 3
Incidence and severity of chronic GVHD
Incidence of nonrelapsing mortality at 100 days and at 1 year after transplantation
Incidence of relapse
Relapse-free survival
Incidence of Epstein-Barr virus activation and post-transplantation lymphoproliferative disease

CONTACTS AND LOCATIONS:
Overall Officials: Paul V. O'Donnell, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States